CLINICAL TRIAL: NCT06406205
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Comparing the Efficacy and Safety of QLG1074 With Placebo in Achieving Renal Remission in Subjects With Active Lupus Nephritis
Brief Title: A Study of QLG1074 Combined With Background Therapy in Subjects With Active Lupus Nephritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLG1074-301
Record Dates: First submitted 2024-03-20; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voclosporin（QL1074） (Experimental): oral, 23.7 mg twice daily (BID)，52 weeks Drug: Voclosporin calcineurin inhibitor Other Names: QL1074
  Interventions: Drug: Voclosporin（QL1074）
- Placebo Oral Capsule (Placebo Comparator): Voclosporin placebo, oral, 3 capsules twice daily (BID)，52 weeks Drug: Placebo Oral Capsule matching placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Voclosporin（QL1074） — QL1074 23.7 mg BlD will be administered as a fixed dose without the use of therapeutic drugmonitoring. The protocol contains provisions for management of dose based on safety concerns, in particular, BP and renal function，can be managed by dose reduction and temporary of QL1074 to interruption.
  Arms: Voclosporin（QL1074）
Drug: Placebo — Placebo softgel capsules, identical to 7.9 mg QL1074, will be provided. The administration plan and dosage management regulations are the same as QL1074.
  Arms: Placebo Oral Capsule

SUMMARY:
The purpose of this study is to assess the efficacy of QL1074 compared with placebo in achieving renal response after 52 weeks of therapy in subjects with Active Lupus Nephritis.

DETAILED DESCRIPTION:
The aim of the current study is to investigate whether QL1074, added to the standard of care treatment in active lupus nephritis (LN), is able to reduce disease activity over a treatment period of 52 weeks. The background therapy will be mycophenolate mofetil (MMF) and initial treatment with IV methylprednisolone, followed by a reducing course of oral corticosteroids. Subjects with active LN will be eligible to enter the study. They are required to have a diagnosis of LN according to established diagnostic criteria and clinical and biopsy features suggestive of active nephritis. Efficacy will be assessed by the ability of the drug combination to reduce the level of proteinuria (as measured by Urine Protein Creatinine Ratio (UPCR)) while demonstrating an acceptable safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent before any study-specific procedures are performed.
2. Male or female subjects with a minimum age of 18 (or legal age of consent if >18 years) to 75 years of age, inclusive, at the time of screening (Visit 1).
3. Previous diagnosis of systemic lupus erythematosus (SLE) according to the American College of Rheumatology criteria (1997)
4. Subjects with evidence of active nephritis, According to the 2018 International Society of Nephrology/Society of Nephropathology (ISN/RPS) classification criteria for lupus nephritis, defined as follows:

   * Kidney biopsy result within 2 years prior to screening indicating Class III, IV (alone or in combination with Class V), or Class V LN, Biopsy results must be reviewed with the Investigator to confirm eligibility.
   * UPCR of a minimum of ≥1.5 mg/mg for Class III/IV or to a minimum of ≥2 mg/mg for Class V at screening.
   * If the subject provides a biopsy report within 2 years but more than 6 months before screening, the UPCR needs to be doubled at least within 6 months before screening.
5. According to the Investigators' evaluation, subject requires high-dose corticosteroids and immunosuppressive therapy.
6. Subject is willing to take oral MMF for the duration of the study, either by continuing current MMF therapy or by initiating it on or before the Baseline Visit.
7. Fertile subjects (both male and female) must agree to use reliable contraception methods with their partners from the time of signing the informed consent form until 3 months after the end of the trial; women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline.

Exclusion Criteria:

1. Estimated glomerular filtration rate (eGFR) as calculated by the Chronic Kidney Disease Epidemiology Collaboration equation of ≤45 mL/minute/1.73 m2 at screening.
2. urrently taking or planning to use drugs or treatments listed in the Prohibited Drugs (Section 5.5) during the trial, including not completing the required washout.
3. Currently requiring renal dialysis (hemodialysis or peritoneal dialysis) or expected to require dialysis during the study period.
4. A previous kidney transplant or planned transplant within study treatment period.
5. Any known hypersensitivity or contraindication to any of the drugs planned to be used (including but not limited to: MMF, Mycophenolate Sodium, Cyclosporine, Voclosporin, Corticosteroids) or any components of these drug products.
6. Current or medical history of:

   * The subject has a history of drug abuse or alcohol abuse within 2 years before the screening period;
   * Malignancy within 5 years of screening, with the exception of basal and squamous cell carcinomas treated by complete excision. Subjects with cervical dysplasia that is cervical intraepithelial neoplasia 1, but have been treated with conization or loop electrosurgical excision procedure and have had a normal repeat Papanicolaou test are allowed;
   * Lymphoproliferative disease or previous total lymphoid irradiation;
   * Severe viral infection (e.g., cytomegalovirus, hepatitis B virus, hepatitis C virus) within 3 months of screening; or known HIV infection. Severe viral infection is defined as active disease requiring antiviral therapy;
   * Active tuberculosis (TB), or known history of TB/evidence of old TB if not taking prophylaxis with isoniazid;
7. Other known clinically significant active medical conditions, such as:

   * Severe cardiovascular disease including congestive heart failure, history of cardiac dysrhythmia, congenital long QT syndrome or Hypertension with poor control (systolic blood pressure ≥165mmHg and/or diastolic blood pressure ≥105mmHg after treatment with 2 or more drugs). QT interval duration corrected for heart rate using method of Fridericia exceeding 480 msec in the presence of a normal QRS interval (<110 msec) at time of screening will result in exclusion;
   * Liver dysfunction (aspartate aminotransferase, alanine aminotransferase, or bilirubin ≥2.5 times the upper limit of normal) at screening and, if abnormal at screening, then confirmed that the levels have returned to <2.5 times upper limit of normal before randomization;
   * Chronic obstructive pulmonary disease or asthma requiring oral steroids;
   * Bone marrow insufficiency unrelated to active SLE (according to Investigator judgment) with white blood cell count <2.5×109/L; absolute neutrophil count <1.3×109/L; thrombocytopenia (platelet count <50×109/L);
   * According to the evaluation of the investigator, the subject suffered from active bleeding;
   * Patients with infections requiring intravenous antibiotic treatment (antibacterial drugs, antiviral drugs, antifungal drugs, or antiparasitic drugs) during screening;
8. According to the researchers' assessment, the subjects have other congenital or acquired immune diseases (except for SLE and LN), for which the condition or the treatment of the condition may affect the study assessments or outcomes (e.g., scleroderma with significant pulmonary hypertension; any condition for which additional immunosuppression is indicated). Overlapping conditions for which the condition or treatment is not expected to affect assessments or outcomes (e.g.,Sjögren's syndrome) are not excluded.
9. No vaccines using live vaccines or attenuated live vaccines are allowed in the 4 weeks before the screening and while taking the study treatment.
10. According to the evaluation of the investigators, there have been significant, unstable or poorly controlled physical/mental illnesses or traumas that may affect the progress or results of the trial within the first 6 months of the screening period.
11. Women who are pregnant or breastfeeding.
12. Participated in another drug or device trial within 4 weeks before the screening period or within 5 half-lives of the drug (whichever is longer).
13. The subject has participated in previous clinical trials of Voclosporin, was randomly assigned to a group, and received treatment with the trial drug.
14. According to the assessment of the investigators, there may be conditions that affect the results of the trial or that the risks to the subjects outweigh the benefits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Complete Renal Remission at Week 52 | Week 52
  The primary efficacy endpoint was the number of subjects showing complete renal response at Week 52. Complete renal response was adjudicated based on blinded data by an independent Clinical Endpoints Committee based on meeting the following criteria： UPCR of ≤0.5 g/g & eGFR ≥60 mL/min/1.73 m2 or no confirmed decrease from baseline in eGFR of >20%

SECONDARY OUTCOMES:
Time to Urine Protein Creatinine Ratio of ≤0.5 g/g(Number of Days) | 52 Weeks
  Time in days to reduction in Urine Protein Creatinine Ratio to decrease to 0.5 g/g or less.
Number of Participants With Reduction in Urine Protein Creatinine Ratio to 0.5 g/g or Less | 52 Weeks
  Number of Participants With Reduction in Urine Protein Creatinine Ratio to 0.5 g/g or Less
Number of Subjects With Partial Renal Response at Week 52 | Week 52
  Number of subjects with partial Renal Response (defined as a 50% reduction in UPCR from baseline) at Week 52. Baseline UPCR is the average of 2 pre-randomisation values.
Time to 50% Reduction in UPCR (Number of Days) | 52 Weeks
  Time in days to reduction in Urine Protein Creatinine Ratio to decrease by 50% compared to baseline. Baseline is the average of two pre-randomisation values.
Number of Subjects With Partial Renal Response at Week 24 | Week 24
  Number of subjects with partial Renal Response (defined as a 50% reduction in UPCR from baseline) at Week 24. Baseline UPCR is the average of 2 pre-randomisation values.
Number of Subjects With Renal Response With Low Dose Steroids | Week 24 and Week 52
  Programmed Renal Response whilst on low dose steroids (<2.5 mg/day) for the preceding 8 Weeks at Weeks 24 and 52
Change From Baseline in UPCR | Baseline and Weeks 2, 4, 8, 12, 16, 16, 20, 24, 30, 36, 42, 48 and 52.
  Change from baseline by visit in Urine Protein Creatinine Ratio. Baseline is the average of two pre-randomisation values.
Proportion of subjects experiencing a confirmed 30% decrease or more fom baseline in eGFR at each timepoint | Baseline and Weeks 2, 4, 8, 12, 16, 16, 20, 24, 30, 36, 42, 48 and 52.
  Number of subjects with a 30% or more decrease in estimated glomerular filtration rate compared to baseline at each visit time point that meets diagnostic criteria.
Change from baseline by visit in Serum Creatinine, Urine Protein, and estimated Glomerular Filtration rate. | Baseline and Weeks 2, 4, 8, 12, 16, 16, 20, 24, 30, 36, 42, 48 and 52.
  Change from baseline by visit in Serum Creatinine, Urine Protein, and estimated Glomerular Filtration rate. eGFR is corrected to a maximum value of 90 mL/min/1.73 m2
Change From Screening in Immunology Parameters (Complement 3 (C3), C4, and Anti-Double-Stranded DNA) | Week 24 and Week 52
  Change from baseline by visit in Immunology Parameters (Complement 3 (C3), C4, and Anti-Double-Stranded DNA). The immunological baseline data is the numerical value during the screening period.
Change From Baseline in Patient Reported Outcomes | Week 12, Week 24 and Week 52
  Health-related quality of life (HRQoL) information was collected using the Short Form Health Survey (SF-36) HRQoL assessment and the LupusPRO (v1.7) assessment.
  The SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. Scoring ranges from 0 to 100 with higher scores reflecting better health.
  LupusPro assessment is a patient-reported questionnaire regarding the effect of lupus or its treatment on the patient's health, quality of life, and the medical care received related to lupus. The questionnaire consists of 43 questions within 8 HRQOL domains and 4 Non-HRQoL domains. Scores range from 0 to 100 with higher scores reflecting better quality of life.
Change From Baseline in Safety of Estrogens in Systemic Lupus Erythematosus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA - SLEDAI) | Week 24 and Week 52
  The SELENA-SLEDAI tool is a cumulative and weighted index used to assess disease activity across 24 different disease descriptors in patients with lupus. A patient's SELENA-SLEDAI total score is the sum of all marked lupus related descriptors (seizure, psychosis, organic brain syndrome, visual disturbance, cranial nerve disorder, lupus headache, cerebrovascular accident, vasculitis, arthritis, myositis, urinary casts, hematuria, proteinuria, pyuria, new rash, alopecia, mucosal ulcers, pleurisy, pericarditis, low complement, increased DNA binding, fever, thrombocytopenia, leukopenia). A total score can fall between 0 and 105, with a higher score representing a more significant degree of disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Guangyan Cai, MD, Study Chair — Chincse PLA General Hosptial
Locations (10):
- China (10):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - The People's Hospital of Bozhou, Bozhou, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Chincse PLA General Hosptial, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi

IPD SHARING:
Plan to Share IPD: No